CLINICAL TRIAL: NCT03944161
Title: Effectiveness and Cost-Effectiveness Study of Medical Nutrition in Malnourished Patients in Spain
Acronym: COSENUT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The COVID-19 pandemic increased hospital pressure and suspended hospital visits, making it impossible to continue with recruitment. The project has been terminated.
Sponsor: Asociación Española de Fabricantes y Distribuidores de Productos de Nutrición Enteral (Other)
Collaborators: WEBER Economía y Salud S.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01_2019
Record Dates: First submitted 2019-04-15; First posted 2019-05-09 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Malnutrition; Nutrition Disorders
Keywords: nutritional supplement; cost-effectiveness; cost-utility
MeSH Terms: conditions — Malnutrition; Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will receive an oral nutrition supplement bottle (200/220 ml) with >20 % of protein and 1.5 Kcal/ml without fibre twice a day during 12 weeks and nutritional advice.
  Interventions: Dietary Supplement: Oral nutrition supplement; Other: Nutritional advice
- Control group (Active Comparator): Participants in the control group will receive nutrition advice
  Interventions: Other: Nutritional advice

INTERVENTIONS:
Dietary Supplement: Oral nutrition supplement — Hypercaloric and high protein supplement
  Arms: Intervention group
Other: Nutritional advice — Advice given by the clinician

SUMMARY:
The present study aims to evaluate the use of oral nutritional supplementation in persons with some clinical conditions presenting malnutrition in some extent.

DETAILED DESCRIPTION:
COSNUT pretends to assess the cost-effectiveness and cost-utility of oral nutritional supplementation (ONS) in persons with malnutrition and other clinical conditions. The effectiveness will be evaluated by comparing the intervention group having ONS vs a control group only with nutrition advice. The effectiveness and resource use will be collected using quality of life assessment tools, body mass index, change in malnutrition state, number of hospital admissions, medical visits...

Unitary costs for Spain will be extracted from databases and official publications and will be applied to the number of resources used in order to calculate the costs in each of the groups. Finally, the incremental cost-effectiveness ratio will be estimated and presented.

ELIGIBILITY:
Inclusion Criteria:

* >18 y
* Nutritional status B or C (GSA criteria)
* Presenting one of the following conditions:
* Cancer patient after surgery, radiotherapy on antineoplastic treatment.
* Hip fracture
* Heart failure NYHA (New York Heart Association) III-IV.
* Breathing failure GOLD 3 o 4: FEV1 (forced expiratory volume at one second ) <50%.
* Renal failure GFR<30 (glomerular filtration rate )
* Participants agreeing the informed consent

Exclusion Criteria:

* Cancer patients: esophagus, stomach, pancreas and Head and neck
* Hospital admitted patients at the time of recruitment
* Life expectancy below 3 months
* Pregnant or nursing women
* Use of oral nutritional supplements in the three months prior the enrolment
* History of allergy to oral nutritional supplements
* Diabetes mellitus type 1.
* Participation in any other study at the time of enrolment
* Cognitive limitations to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Body mass index | baseline
  Index for relating weight to height. Abbreviated BMI. BMI is a person's weight in kilograms (kg) divided by his or her height in meters squared
Body mass index | 12 weeks
  Index for relating weight to height. Abbreviated BMI. BMI is a person's weight in kilograms (kg) divided by his or her height in meters squared
Body mass index | 6 months
  Index for relating weight to height. Abbreviated BMI. BMI is a person's weight in kilograms (kg) divided by his or her height in meters squared
Change in nutritional status | from baseline-12 weeks
  Change in the Global Subjective Assessment (this scale categorize participants into A, B or C being A the best nutritional status and C the worst.)
Change in nutritional status | from basal-6 months
  Change in the Global Subjective Assessment (this scale categorize participants into A, B or C being A the best nutritional status and C the worst.)
Number of participants Diagnosed of malnutrition | from baseline-12 weeks
  Diagnosis of malnutrition using GLIM criteria
Number of participants Diagnosed of malnutrition | from baseline-6 months
  Diagnosis of malnutrition using GLIM criteria
Health related quality of life | from baseline-12 weeks
  EuroQoL 5 dimensions and 5 levels(EQ5D5L) (scale between 0 which is the death and 1 which is the best health status)
Health related quality of life | from baseline-6 months
  EuroQoL 5 dimensions and 5 levels(EQ5D5L) (scale between 0 which is the death and 1 which is the best health status)
Functional status | from baseline-12 weeks
  Katz index (this index categorize in one of 7 categories: A,B,C,D,E,F,G from independent for all functions (A) to dependent for all functions (G))
Functional status | from baseline-6 months
  Katz index (this index categorize in one of 7 categories: A,B,C,D,E,F,G from independent for all functions (A) to dependent for all functions (G))
Strength and endurance | from baseline-12 weeks
  30-second Chair Stand Test
Strength and endurance | from baseline-6 months
  30-second Chair Stand Test
Strength | from baseline-12 weeks
  hand grip strength test
Strength | from baseline-6 months
  hand grip strength test
Number of Hospital admittance | at 30 days
  Number of admittance from randomization
Number of Hospital admittances | from randomization to 6 months
  Number of admittance from randomization
Number of Medical doctor visits | from randomization to 6 months
  Visits to any outpatient medical office

SECONDARY OUTCOMES:
Number of deaths | from randomization to 6 months
  mortality registry
Number of Infections | at 6 months
  Any diagnosed infection by a medical doctor
Number of secondary effects related to the intervention | from randomization to 6 months
  Any undesirable effect due to the intervention

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Complejo Hospitalario Regional Reina Sofía, Córdoba, Andalusia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Aragon
  - Complejo Asistencial Universitario de León, León, Castille and León
  - Complejo Asistencial de Segovia, Segovia, Castille and León
  - Hospital Universitari Germans Trias I Pujol de Badalona, Badalona, Catalonia
  - Hospital Universitari Joan Xxiii de Tarragona, Tarragona, Catalonia
  - Hospital General Nuestra Señora Del Prado, Talavera de la Reina, Toledo

IPD SHARING:
Plan to Share IPD: No